CLINICAL TRIAL: NCT00119262
Title: Phase II Feasibility Trial Incorporating Bevacizumab Into Dose Dense Doxorubicin and Cyclophosphamide Followed by Paclitaxel in Patients With Lymph Node Positive Breast Cancer
Brief Title: Bevacizumab and Combination Chemotherapy in Patients With Lymph Node Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02977; NCI-2012-02977 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH); E2104 (Other: Eastern Cooperative Oncology Group); E2104 (Other: CTEP)
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Results first posted 2011-04-28 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-12

CONDITIONS: Male Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Bevacizumab; Paclitaxel; Taxes; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Radiotherapy; Radiation; Tamoxifen; Aromatase Inhibitors

ARMS (2):
- Arm I (combination chemotherapy, 18 courses of bevacizumab) (Experimental): See detailed description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: bevacizumab; Drug: paclitaxel; Biological: filgrastim; Biological: pegfilgrastim; Radiation: radiation therapy; Drug: tamoxifen citrate; Drug: aromatase inhibition therapy
- Arm II (combination chemotherapy, 22 courses of bevacizumab) (Active Comparator): See detailed description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: bevacizumab; Drug: paclitaxel; Biological: filgrastim; Biological: pegfilgrastim; Radiation: radiation therapy; Drug: tamoxifen citrate; Drug: aromatase inhibition therapy

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: tamoxifen citrate — Given orally
  Other Names: Nolvadex; TAM; tamoxifen; TMX
Drug: aromatase inhibition therapy — Receive aromatase inhibition therapy
  Other Names: inhibition therapy, aromatase

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with combination chemotherapy works in treating patients who have undergone surgery for breast cancer that has spread to the lymph nodes. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with more than one chemotherapy drug (combination chemotherapy), may be a better way to block tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the incidence of clinically apparent cardiac dysfunction in patients with lymph node positive breast cancer treated with bevacizumab and dose dense doxorubicin/cyclophosphamide followed by paclitaxel (ddAC > T).

SECONDARY OBJECTIVES:

I. To evaluate changes in LVEF during treatment. II. To evaluate non-cardiac toxicity.

OUTLINE: This is a non-randomized, multicenter study. Patients are sequentially assigned to 1 of 2 treatment arms.

Arm A: Patients receive doxorubicin IV, cyclophosphamide IV over 20-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SQ) on days 2-11 or pegfilgrastim SC on day 2. Treatment repeats every 14 days for 4 courses. Patients then receive paclitaxel IV over 3 hours and bevacizumab IV over 30-90 minutes on day 1. Patients also receive G-CSF or pegfilgrastim as above. Treatment with paclitaxel, bevacizumab, and G-CSF or pegfilgrastim repeats every 14 days for 4 courses. Patients then receive bevacizumab alone every 14 days for up to 18 courses.

Arm B: Patients receive doxorubicin, cyclophosphamide, and G-CSF or pegfilgrastim as in group I. Patients then receive paclitaxel, bevacizumab, and G-CSF or pegfilgrastim as in group I. Patients then receive bevacizumab alone every 14 days for up to 22 courses.

Treatment in both groups continues in the absence of disease recurrence or unacceptable toxicity.

Patients who require radiotherapy (post-lumpectomy) or who plan radiotherapy at the discretion of the investigator (post-mastectomy) undergo radiotherapy beginning within 6 weeks after the completion of chemotherapy.

Premenopausal patients with estrogen receptor (ER) and/or progesterone receptor (PR) positive disease receive oral tamoxifen once daily for 5 years beginning at the time of radiotherapy or within 6 weeks after the completion of chemotherapy. Postmenopausal patients with ER and/or PR positive disease receive an aromatase inhibitor (e.g., anastrozole, letrozole, or exemestane) or tamoxifen followed by an aromatase inhibitor once daily for up to 10 years.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for up to 3 years from study entry.

ACCRUAL: A total of 226 patients (104 on arm A and 122 on arm B) were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast with involvement of at least one axillary or internal mammary lymph node on routine histologic examination with hematoxylin and eosin staining; NOTE: patients with axillary or internal mammary node involvement only demonstrated by immunohistochemistry are not eligible
* Patients must have completed definitive breast surgery including total mastectomy and axillary dissection (modified radical mastectomy), total mastectomy and sentinel node biopsy, lumpectomy and axillary dissection, or lumpectomy and sentinel node biopsy; NOTE: axillary dissection is strongly encouraged in patients with lymph node involvement identified on sentinel node biopsy
* Margins of lumpectomy or mastectomy must be histologically free of invasive breast cancer and ductal carcinoma in situ (DCIS); patients with resection margins positive for lobular carcinoma in situ (LCIS) are eligible
* (ARM A ONLY) Interval between last surgery for breast cancer (lumpectomy, mastectomy, sentinel node biopsy, axillary dissection or re-excision of lumpectomy margins) and D1 must be > 28 days and =< 84 days
* ECOG performance status of 0-2
* Absolute neutrophil count >= 1000/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 mg/dL
* AST =< 2 upper limit of normal
* Serum creatinine =< 1.5 mg/dL
* Urine protein: creatinine ratio < 1.0
* PT INR =< 1.5
* PTT =< 1.5 x normal
* LVEF >= institutional limits of normal by MUGA or ECHO
* Prior to registration the investigator must specify if radiation is planned; patients who have undergone a lumpectomy must receive radiation; post-mastectomy radiation is at the investigator's discretion
* Patients with HER2+ (3+ by IHC or FISH+) breast cancer are not eligible and should be treated with a trastuzumab-based adjuvant therapy
* Patients with synchronous bilateral breast cancer (diagnosed within one month) are eligible if the higher TMN stage tumor meets the eligibility criteria for this trial
* Patients must not have clinical evidence of inflammatory disease or fixed axillary nodes (N2) at diagnosis
* Patients must not have received prior cytotoxic chemotherapy, hormonal therapy or radiation for this breast cancer; prior treatment with an anthracycline, anthracenedione or taxane for any condition is not allowed; NOTE: prior use of tamoxifen for chemoprevention is allowed but must be discontinued at study entry; similarly prior raloxifene use is allowed but must be discontinued at study entry
* Patients must not have had a major surgical procedure within 4 weeks of entry; NOTE: non-operative biopsy or placement of a vascular access device is not considered a major surgery
* Patients must not have clinically significant cardiovascular disease including:

  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Grade II or greater peripheral vascular disease
  * Uncontrolled hypertension defined as SBP > 160 or DBP > 90
  * Any prior history of cerebrovascular disease including TIA or stroke
* Patients must not require therapeutic anticoagulation; patients with a history of deep venous thrombosis or pulmonary embolism are not eligible; NOTE: prophylactic use of anticoagulants to maintain patency of a vascular assess device is permitted
* Patients may not require regular use of aspirin (daily for >= 10 days at doses of > 325 mg/day) or regular therapeutic doses of other nonsteroidal anti-inflammatory agents known to inhibit platelet function; additionally, patients using any of the following drugs known to inhibit platelet function are not eligible: dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and cilostazol (Pletal); NOTE: regular use of Cox-2 inhibitors is permitted; NOTE: low-dose aspirin is permitted
* Patients must not have a non-healing wound or fracture; patients with an abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months are excluded
* Patients must not have hypersensitivity to paclitaxel or drugs using the vehicle Cremophor, Chinese hamster ovary cell products or other recombinant human antibodies
* Patients who have experienced myocardial infarction or unstable angina within 12 months are excluded
* Patients who have had experienced an arterial thrombotic event within 12 months are excluded
* Patients must not have uncontrolled or clinical significant arrhythmia
* Women must not be pregnant or breast-feeding due to the potential harmful effects of bevacizumab on the developing fetus; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males are required to use an accepted and effective method of contraception while on study and for at least 3-4 months after the last dose of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2005-10; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E2104 was opened on October 6,2005, and closed on November 6, 2006 with the final accrual of 226 patients.Study participants included Eastern Cooperative Oncology Group (ECOG) entire group, North Central Cancer Treatment Group (NCCTG) entire group and Cancer and Leukemia Group B (CALGB) entire group.
Groups:
- Arm A (ddBAC > BT > B): Dose dense bevacizumab, cyclophosphamide and doxorubicin, followed by paclitaxel and bevacizumab, followed by bevacizumab
- Arm B (ddAC > BT > B): Dose dense doxorubicin and cyclophosphamide, followed by paclitaxel and bevacizumab, followed by bevacizumab
Period: Overall Study
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B)
Started | 104 | 122
Eligible | 103 | 120
Treated | 103 | 120
Eligible and Treated | 102 | 119
Completed | 58 | 64
Not Completed | 46 | 58
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Adverse Event | 33 | 35
Not completed — other disease | 0 | 2
Not completed — ineligble | 1 | 2
Not completed — others | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B) | Total
Number analyzed (Participants) | 103 | 120 | 223
Age, Continuous [Median (Full Range); unit: years] | 50 [33 to 76] | 50 [27 to 76] | 50 [27 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 119 | 222
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 103 | 120 | 223

OUTCOME MEASURES:

1. Primary Outcome: Congestive Heart Failure Rate
Description: Clinical congestive heart failure includes patients with symptomatic decline in LVEF to at or below the lower limit of normal (LLN), or symptomatic diastolic dysfunction. 223 treated patients were included in the analysis.
Time Frame: assessed on day 1 of cycles 5, 9, 17 and 25, and at end of treatment, then every 3 months for <2 years and every 6 months for 2-3 years from study entry
Population: 223 treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B)
Number analyzed (Participants) | 103 | 120
percentage of participants | 2.9 [0.6 to 8.3] | 2.5 [0.5 to 7.1]

2. Secondary Outcome: Proportion of Patients With Absolute Decrease in Left Ventricular Ejection Fraction (LVEF) Levels Post Doxorubicin and Cyclophosphamide(AC)
Description: The endpoint was measured by absolute decrease from baseline in LVEF of >15% or >10% decline from baseline to below the LLN post doxorubicin and cyclophosphamide (AC) Day 1 Cycle 5 (DIC5). 207 patients who were treated and had baseline and DIC5 LVEF values were included in the analysis.
Time Frame: assessed on day 1 of cycles 5, 9, 17, 25, and at end of treatment
Population: Patients who were treated and had baseline and DIC5 LVEF values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B)
Number analyzed (Participants) | 94 | 113
percentage of participants | 7.4 [3.0 to 14.7] | 3.5 [0.9 to 8.8]
Statistical Analysis 1: Comparison: Arm A (ddBAC > BT > B) vs Arm B (ddAC > BT > B); Test type: Superiority or Other; p = 0.12, Fisher Exact

3. Secondary Outcome: Proportion of Patients With Absolute Decrease in LVEF Levels Post Bevacizumab
Description: The endpoint was measured by absolute decrease from baseline in LVEF of >15% or >10% decline from baseline to below the LLN post bevacizumab (the end of treatment). 158 patients who were treated and had baseline and end of treatment LVEF values were included in the analysis.
Time Frame: assessed on day 1 of cycles 5, 9, 17, 25, and at end of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B)
Number analyzed (Participants) | 72 | 86
percentage of participants | 15.3 [7.9 to 25.7] | 11.6 [5.7 to 20.3]
Statistical Analysis 1: Comparison: Arm A (ddBAC > BT > B) vs Arm B (ddAC > BT > B); Test type: Superiority or Other; p = 0.32, Fisher Exact

ADVERSE EVENTS:
Time Frame: assessed at the end of each cycle while on treatment and for 30 days after the end of treatment, and assessed every 3 months if patient is <2 years and every 6 months if patient is 2-3 years from study entry
Arm/Group | Arm A (ddBAC > BT > B) | Arm B (ddAC > BT > B)
Serious Adverse Events (participants affected / at risk) | 71/103 | 65/120
Other Adverse Events (participants affected / at risk) | 103/103 | 120/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (ddBAC > BT > B) (N=103) | Arm B (ddAC > BT > B) (N=120)
Allergic reaction (Immune system disorders) | 4 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 4
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Investigations) | 22 | 27
Neutropenia (Investigations) | 28 | 31
Thrombocytopenia (Investigations) | 2 | 2
Cardiac-Ischemia (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 13 | 13
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 4 | 4
Fatigue (General disorders) | 11 | 7
Fever w/o neutropenia (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 1
Hot flashes (Vascular disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 0
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 3 | 3
Muco/stomatitis (symptom), pharynx (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Rectum, hemorrhage (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5
Infection w/gr3-4 neut,lung (Infections and infestations) | 1 | 0
Infection w/gr3-4 neut, mucosa (Infections and infestations) | 0 | 1
Infection w/gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0
Infection w/gr0-2 neut, bronchus (Infections and infestations) | 1 | 0
Infection w/gr0-2 neut, catheter (Infections and infestations) | 1 | 0
Infection w/gr 0-2 neut, lung (Infections and infestations) | 1 | 0
Infection w/gr 0-2 neut, pharynx (Infections and infestations) | 0 | 1
Infection w/gr 0-2 neut, skin (Infections and infestations) | 1 | 2
Infection w/gr 0-2 neut, urinary tract (Infections and infestations) | 1 | 0
Infection w/ unknown ANC, mucosa (Infections and infestations) | 0 | 1
Infection w/ unknown ANC, oral activity/gums (Infections and infestations) | 0 | 1
Infection w/ unknown ANC, upper airway NOS (Infections and infestations) | 1 | 0
Infection w/gr 0-2 neut, blood (Infections and infestations) | 1 | 0
ALT increased (Hepatobiliary disorders) | 2 | 1
Amylase increased (Investigations) | 1 | 0
AST increased (Hepatobiliary disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Nonneuropathic generalized weakness (General disorders) | 1 | 0
CNS cerebrovascular Ischemia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 8 | 10
Syncope (Nervous system disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gallbladder, pain (Hepatobiliary disorders) | 1 | 0
Head/headache (Nervous system disorders) | 1 | 8
Joint,pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Muscle,pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Neuropathic,pain (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 0 | 4
Vascular assess, Thrombosis/Embolism (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 2
Lymphopenia (Investigations) | 3 | 9
Proteinuria (Renal and urinary disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (ddBAC > BT > B) (N=103) | Arm B (ddAC > BT > B) (N=120)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Anemia (Blood and lymphatic system disorders) | 51 | 60
Leukopenia (Investigations) | 42 | 41
Lymphopenia (Investigations) | 5 | 12
Neutropenia (Investigations) | 28 | 19
Thrombocytopenia (Investigations) | 25 | 32
Hypertension (Vascular disorders) | 45 | 43
Left ventricular systolic dysfunction (Cardiac disorders) | 19 | 20
Fatigue (General disorders) | 86 | 102
Fever w/o neutropenia (General disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 19 | 24
Rigors/chills (General disorders) | 8 | 15
Sweating (General disorders) | 8 | 16
Weight gain (Investigations) | 12 | 14
Weight loss (Investigations) | 32 | 36
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 93 | 91
Nail change (Skin and subcutaneous tissue disorders) | 17 | 28
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 35 | 31
Radiation dermatitis (Injury, poisoning and procedural complications) | 7 | 6
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 12 | 9
Hot flashes (Vascular disorders) | 24 | 43
Anorexia (Metabolism and nutrition disorders) | 43 | 43
Constipation (Gastrointestinal disorders) | 36 | 50
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 37 | 46
Dry mouth (Gastrointestinal disorders) | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 36 | 43
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 63 | 62
Muco/stomatitis (symptom), pharynx (Gastrointestinal disorders) | 15 | 12
Nausea (Gastrointestinal disorders) | 88 | 100
Taste disturbance (Gastrointestinal disorders) | 26 | 37
Vomiting (Gastrointestinal disorders) | 38 | 40
Oral activity, hemorrhage (Gastrointestinal disorders) | 7 | 9
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 6 | 3
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 39 | 35
Edema limb (General disorders) | 5 | 13
Alkaline phosphatase increased (Investigations) | 36 | 37
ALT increased (Hepatobiliary disorders) | 25 | 23
AST increased (Hepatobiliary disorders) | 18 | 33
Bilirubin increased (Investigations) | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 9
Hemoglobinuria (Renal and urinary disorders) | 3 | 6
Hypokalemia (Metabolism and nutrition disorders) | 5 | 11
Proteinuria (Renal and urinary disorders) | 11 | 23
Hyponatremia (Metabolism and nutrition disorders) | 6 | 6
Dizziness (Nervous system disorders) | 9 | 18
Anxiety (Psychiatric disorders) | 17 | 5
Depression (Psychiatric disorders) | 9 | 12
Neuropathy-motor (Nervous system disorders) | 7 | 9
Neuropathy-sensory (Nervous system disorders) | 72 | 89
Vision-blurred (Eye disorders) | 2 | 8
Tearing (Eye disorders) | 6 | 14
Ocular-other (Eye disorders) | 6 | 2
Abonominal pain (Gastrointestinal disorders) | 6 | 6
Back, pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 20
Chest/thoracic pain NOS (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Extremity-limb,pain (Musculoskeletal and connective tissue disorders) | 4 | 9
Head/headache (Nervous system disorders) | 39 | 51
Joint,pain (Musculoskeletal and connective tissue disorders) | 63 | 75
Muscle,pain (Musculoskeletal and connective tissue disorders) | 57 | 76
Pain NOS (Gastrointestinal disorders) | 6 | 3
Pain-other (General disorders) | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 30
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Irregular menses (Reproductive system and breast disorders) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less